CLINICAL TRIAL: NCT02844491
Title: Study of T Specific Immune Response Against Delta-CD20 Peptide in Hematological Malignancies B
Acronym: Epitopes-LNH01
Status: Terminated | Type: Observational
Why Stopped: Difficulty of recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2012/157
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hematological Malignancies B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood samples will be realized at inclusion and Peripheral Blood Mononuclear Cells (PBMC) will be collected.
  * Tumor tissues will be collected if available.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: In Cohort A, patients will be included either in the group "sustainable response"or in the "short / refractory response" group.
  - "sustainable response" group : patient with NHL diffuse large B cells, and persistent complete response for at least 6 months after first-line treatment with Rituximab OR patient with follicular NHL, mantle NHL, NHL marginal zone or Waldenstrom's disease in complete response or partial stable response for at least 1 year after first line treatment with Rituximab
  "short / refractory response" group : patient with NHL diffuse large B cells, refractory or relapsed in less than 6 months after at least one line of treatment with Rituximab OR patient with follicular NHL, mantle NHL, NHL marginal zone or Waldenstrom's disease refractory or relapsed / progression within less than 1 year after at least one line of treatment with Rituximab
  Interventions: Other: additional biological samples
- Cohort B: For Cohort B patients will be included either in the group "B hematologic therapeutic abstention" or in the group "any blood disease not treated with anti-CD20 antibodies."
  "B hematologic therapeutic abstention" group : patient with hematological malignancy whatever the initial expansion stage
  "any blood disease not treated with anti-CD20 antibodies" group : patient with follicular NHL, mantle NHL, NHL marginal zone or Waldenstorm disease without treatment criteria at diagnosis and with stable disease for at least 6 months
  Interventions: Other: additional biological samples

INTERVENTIONS:
Other: additional biological samples — blood and tissue samples

SUMMARY:
Cancer-specific splice variants gain significant interest as they generate neo-antigens, that could be targeted by immune cells. CD20, a membrane antigen broadly expressed in mature B cell lymphomas, is subject to an alternative splicing named Delta-CD20 leading to loss of membrane expression of the spliced isoform.

The investigators group would now determine if it's possible, in patients with lymphoproliferative B, to detect the presence of a specific memory response to delta-CD20 peptides.

If this memory response exists, it will confirm the interest of this antigen as a target for tumor immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* For all patient :

  •Written informed consent
* For Cohort A :

  * Patient with hematological malignancy of high grade phenotype B (non Hodgkin's lymphoma diffuse large cell) or low grade (mantle cell lymphoma, follicular lymphoma, marginal zone lymphoma or Waldenstrom disease), regardless the initial extension stage.
  * Histologically or cytologically and immunophenotypical confirmed
  * Patient candidate to a second-line or more therapy
  * First-line treatment with rituximab
* For Cohort B :

  * Absence of prior treatment with an anti-CD20 antibody
  * Histologically or cytologically and immunophenotypical confirmed

Exclusion Criteria:

* For all patients :

  * Patient with any medical or psychiatric condition or disease,
  * Patient under guardianship, curatorship or under the protection of justice and pregnant women
* For Cohort A :

  * Patient with chronic lymphocytic leukemia
  * Patient with indolent lymphoma relapsed more than 1 year after treatment with Rituximab
  * Patient allogeneic hematopoietic cells
  * Patient with linked lymphoproliferative syndrome with congenital immunosuppression (eg SCID, XLP ...) or acquired (post-transplant lymphoma)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients studied will be carrying a malignant lymphoproliferative B high grade or low grade treated with an anti-CD20 antibody (cohort A) or hematological whatever type not treated with an anti-CD20 antibody ( cohort B).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-01-22 (Actual); Primary Completion 2014-09-19 (Actual); Study Completion 2014-09-19 (Actual)

PRIMARY OUTCOMES:
presence of Delta-CD20 T cell responses measured by ELISPOT assay | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Besançon, Besançon, France

REFERENCES:
- [Background] Vauchy C, Gamonet C, Ferrand C, Daguindau E, Galaine J, Beziaud L, Chauchet A, Henry Dunand CJ, Deschamps M, Rohrlich PS, Borg C, Adotevi O, Godet Y. CD20 alternative splicing isoform generates immunogenic CD4 helper T epitopes. Int J Cancer. 2015 Jul 1;137(1):116-26. doi: 10.1002/ijc.29366. Epub 2014 Dec 12. PMID 25449106